CLINICAL TRIAL: NCT01531712
Title: Phase II Study of Neoadjuvant Treatment With Gemcitabine, Tarceva and Oxaliplatin Followed by Chemotherapy With Tarceva and Gemcitabine in Patients With Pancreas Adenocarcinoma With Borderline Resectability.
Brief Title: Study of Neoadjuvant Treatment in Patients With Pancreatic Cancer That is Potentially Resectable
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a low recruitment rate since start of recruitment period.
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-20431; 2010-021872-27 (EudraCT Number); GEMERLOXA (Other: ICO)
Record Dates: First submitted 2012-01-11; First posted 2012-02-13 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer
Keywords: neoadjuvant treatment; borderline resectability
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy; Erlotinib Hydrochloride; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QT + QRT (Experimental): Chemotherapy (6 cycles x 14 days): Gemcitabine 1000 mg/m2 (day 1) + Oxaliplatin 100 mg/m2 (day 2) + Tarceva 100 mg/day.
  Chemoradiotherapy (5,5 weeks): Gemcitabine 40 mg/m2 (2 days/week) + Tarceva 100 mg/day + Radiotherapy (1,8 Gy/day x 28 doses, total dose: 50,4 Gy).
  Interventions: Drug: Gemcitabine; Radiation: Radiotherapy; Drug: Tarceva; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 / / 40mg/m2
  Other Names: gemzar
Radiation: Radiotherapy — 50.4 Gy
Drug: Tarceva — 100mg/day
  Other Names: Erlotinib
Drug: Oxaliplatin — 100mg/m2 (only in QT)
  Other Names: ELOXATIN

SUMMARY:
Phase II study of neoadjuvant treatment with Gemcitabine, Tarceva and Oxaliplatin followed by chemotherapy with Tarceva and Gemcitabine in patients with pancreatic adenocarcinoma with borderline resectability. The primary objective is to determine the resectability rate of patients with pancreas adenocarcinoma with borderline resectability determined radiologically, treated with Gemcitabine, Tarceva and Oxaliplatin followed by radiotherapy with Gemcitabine and Tarceva.

DETAILED DESCRIPTION:
Patients with borderline resectable pancreatic adenocarcinoma are more likely to develop perioperative complications due to the complexity of surgery. In these patients there is also an increased risk of systemic relapse due to the advanced stage of the tumor as well as a higher possibility of having positive margins. Therefore, the treatment of these patients need to be decided based on a multidisciplinary strategy. Besides of that the use of systemic neoadjuvant chemotherapy as induction therapy, followed by sequential chemoradiotherapy is a very attractive therapeutic modality.

The neoadjuvant treatment offers the potential advantages of reducing the tumor stage, increasing resectability and decreasing postoperative complications.

The administration of chemotherapy and radiotherapy before surgery represent an strategy for early treatment of micrometastatic disease, present in most of these patients, and to identify patients with rapid progression of the disease.

For all the reasons above, the investigators consider it's of great interest to design new studies that combine systemic neoadjuvant chemotherapy followed by chemoradiotherapy with neoadjuvant intention in patients with pancreas cancer locally advanced.

ELIGIBILITY:
Inclusion Criteria:

* Before the beginning of the specific protocol procedures must be obtained and documented a written consent form. Patients must have sufficient capacity to understand and sign the consent form.
* Exocrine pancreatic potentially resectable carcinoma, histologically confirmed.
* Aged 18-75 years.
* OMS functional state (FE) from 0-2 and Karnofsky functional state 70%.
* Radiologically or measurable disease, defined as borderline resectability disease.
* Appropriate biological parameters: neutrophils > 1.500/mL; platelets > 100.000/mL; hemoglobin > 10 g/dl.Serum creatinine < 1,5 x upper limit of normal (LSN); alkaline phosphatase < 3 x LSN and bilirubin < 1,5 x LSN; AST and ALT 2,5 x LSN.
* Controlled biliary obstruction in all the patients before their inclusion in the study.
* Absence of peripheral neuropathy grade 2.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Previous administration of chemotherapy, radiotherapy or any investigational agents for pancreatic cancer treatment.
* Administration of other experimental treatment during this study or in the previous 6 months.
* Pregnancy, inappropriate or unsafe use of contraceptive methods or women who are breast-feeding.
* Clinically significant heart disease(for example: congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not properly controlled with medication or myocardial infarction in the last 12 months).
* Presence of significant ophthalmologic anomaly, included: severe dry eye syndrome, Sjogren syndrome, dry keratoconjunctivitis, severe exposure keratopathy, conditions that might increase the risk of epithelium complications.
* Patients with lack of physical integrity of the upper gastrointestinal tract or bad absorption syndromes or unable to ingest the tablets.
* Other previous bad or concurrent diseases, with the exception of nonmelanoma skin cancer.
* Medical or psychiatric pathologies that are severe or uncontrolled.
* Distant metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Resectability rate after neoadjuvant treatment with chemotherapy plus chemoradiotherapy. | Two years
  Determine the resectability rate of subjects with borderline resectable pancreatic cancer (radiologically measured) that were treated with Gemcitabine, Tarceva and Oxaliplatin followed by chemoradiotherapy with Gemcitabine and Tarceva.

SECONDARY OUTCOMES:
Median overall survival. | Two years
  To determine the overall survival (OS) and the tumor recurrence pattern (local versus distant).
Rate of resections with engative margins and complete pathological response. | Two years
  To determine the rate of negative margin resections and complete pathological response (cPR).
Response rate to neoadjuvant treatment of tumor markers (CEA, CA19-9) | Two years
  To determine the reponse rate to the neoadjuvant treatment of speficic tumor markers (CEA, Ca19-9).
Ratio of objective responses (RECIST). | Two years
  To determine the ratio of objective responses according to RECIST criteria.
Prognosis accuracy of serum protein profiles | Two years
  To determine the prognosis accuracy of serum protein profiles in these subjects.
Viability of the collection of pre-treatment tumor samples | Two years
  To determine the feasibility of the collection of pre-treatment (baseline) tumor samples and to set pathological correlations with the response after neoadyuvant treatment.
Adverse events | Two years
  To determine the safety, toxicity and feasibility of this therapeutical regimen as neoadyuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Berta Laquente, MD, Principal Investigator — ICO
Locations (1):
- Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain